CLINICAL TRIAL: NCT01504139
Title: The Luteal Phase After GnRHa Trigger - a Proof of Concept Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Helle Olesen Elbaek, Clinical Director, M.D., Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110289
Record Dates: First submitted 2011-12-28; First posted 2012-01-05 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Progesterone Levels; Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Luteal Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- hCG in the late follicular phase + luteal phase (Experimental)
  Interventions: Drug: hCG(r-hCG, Ovitrelle, Merck-Serono, Hellerup, Denmark) in the late follicular phase + luteal phase
- hCG in the follicular phase + luteal phase (Experimental)
  Interventions: Drug: hCG(r-hCG, Ovitrelle,Merck-Serono, Hellerup, Denmark) in the follicular phase + luteal phase
- LH in the luteal phase (Experimental)
  Interventions: Drug: LH(r-LH,Luveris, Merck-Serono, Hellerup, Denmark) in the luteal phase
- vaginal progesterone and estradiol in the luteal phase (Active Comparator)
  Interventions: Drug: vaginal progesterone(Crinone; Merck-Serono, Hellerup, Denmark) and estradiol(Estrofem; Novo Nordisk, Copenhagen, Denmark) in the luteal phase

INTERVENTIONS:
Drug: hCG(r-hCG, Ovitrelle, Merck-Serono, Hellerup, Denmark) in the late follicular phase + luteal phase — when the follicles are over 12 mm FSH(r-hFSH; Gonal-F, Merck-Serono, Hellerup, Denmark) is replaced by hCG (r-hCG, Ovitrelle,Merck-Serono, Hellerup,Denmark).
  Arms: hCG in the late follicular phase + luteal phase
Drug: hCG(r-hCG, Ovitrelle,Merck-Serono, Hellerup, Denmark) in the follicular phase + luteal phase — hCG(r-hCG,Ovitrelle,Merck-Serono, Hellerup, Denmark) is given together with FSH(r-hFSH; Gonal-F, Merck-Serono, Hellerup, Denmark) from the beginning of the FSH(r-hFSH; Gonal-F, Merck-Serono, Hellerup, Denmark)stimulation.
  Arms: hCG in the follicular phase + luteal phase
Drug: LH(r-LH,Luveris, Merck-Serono, Hellerup, Denmark) in the luteal phase — LH(r-LH, Luveris, Merck-Serono, Hellerup, Denmark) replaces progesterone and estradiol in the luteal phase.
  Arms: LH in the luteal phase
Drug: vaginal progesterone(Crinone; Merck-Serono, Hellerup, Denmark) and estradiol(Estrofem; Novo Nordisk, Copenhagen, Denmark) in the luteal phase — The usual dose of vaginal progesterone(Crinone; Merck-Serono, Hellerup, Denmark) and estradiol (Estrofem; Novo Nordisk, Copenhagen, Denmark) is given in the luteal phase-
  Arms: vaginal progesterone and estradiol in the luteal phase

SUMMARY:
The purpose of this study is to investigate levels of progesterone in the luteal phase after various stimulations in the follicular phase and treatment with GnRH antagonist protocol followed by GnRHagonist as induction of ovulation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate levels of progesterone in the luteal phase after various stimulations in the follicular phase and treatment with GnRH antagonist protocol followed by GnRHagonist as induction of ovulation. Furthermore the aim is to explore whether the luteal phase can be supported with small daily boluses of hCG without the administration of exogenous P, while maintaining good reproductive outcome.

ELIGIBILITY:
Inclusion Criteria:

* women from the age of 25 up to 40
* Serum-FSH and serum-LH levels under 12 IU/L
* Length of period between 25 and 34 days
* BMI between 18 and 30

Exclusion Criteria:

* less than 2 ovaries
* uterine abnormalities
* PCOS or UL-PCO (more than 11 follicles over 12 mm in 1 ovary

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Levels of progesterone in the mid-luteal phase. | up to 1-1½years.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Olesen Elbaek, Study Director — The Fertility Clinic, Skive Regional Hospital, Denmark
Locations (1):
- the Fertility clinic, Regional Hospital Skive, Skive, Central Jutland, Denmark

REFERENCES:
- [Derived] Andersen CY, Elbaek HO, Alsbjerg B, Laursen RJ, Povlsen BB, Thomsen L, Humaidan P. Daily low-dose hCG stimulation during the luteal phase combined with GnRHa triggered IVF cycles without exogenous progesterone: a proof of concept trial. Hum Reprod. 2015 Oct;30(10):2387-95. doi: 10.1093/humrep/dev184. Epub 2015 Jul 23. PMID 26209535